CLINICAL TRIAL: NCT00458107
Title: An Ascending Multiple Dose Study of the Safety, Pharmacokinetics, and Pharmacodynamics of SCA-136 Administered Orally to Healthy Japanese and Non-Japanese Female Subjects
Brief Title: Study Evaluating the Safety and Tolerability of SCA-136 in Healthy Japanese and Non-Japanese Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3153A1-1115
Record Dates: First submitted 2007-04-05; First posted 2007-04-09 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Schizophrenia
Keywords: Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Drug: SCA-136

SUMMARY:
This study is being conducted to evaluate the safety and tolerability of ascending multiple oral doses of SCA-136 adminstered to healthy Japanese and non-Japanese female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese women or non-Japanese of child bearing potential using nonhormonal contraceptives.
* Japanese female subjects are defined as being born in Japan but living outside of Japan for less than 5 years.

Exclusion Criteria:

* Any significant disease.
* Positive urine drug screen, increased liver funtion tests, use of prescription drugs.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2007-04; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Adverse events, safety laboratories results, vital signs, and ECGs will be used to monitor subject safety.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Glendale, California, United States